CLINICAL TRIAL: NCT01391936
Title: A Prospective Randomised Trial of Plate Fixation Versus Tension Band Wire for Olecranon Fractures
Brief Title: A Trial of Plate Fixation Versus Tension Band Wire for Olecranon Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andrew D Duckworth (Other)
Responsible Party: Sponsor-Investigator, Andrew D Duckworth, StR, Royal Infirmary of Edinburgh
Organization: Royal Infirmary of Edinburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/RlOST/04
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Displaced Olecranon Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tension Band Wiring (Other): Patients in this arm will receive the tension band wiring technique for fixation of their olecranon fracture.
  Interventions: Procedure: Tension Band Wiring
- Plate fixation (Other): Patients in this arm will receive plate and screw fixation of their olecranon fracture.
  Interventions: Procedure: Plate fixation

INTERVENTIONS:
Procedure: Tension Band Wiring — AO technique of TBW for fixation of fracture.
  Arms: Tension Band Wiring
Procedure: Plate fixation — Patients in this arm will receive plate and screw fixation of their olecranon fracture.
  Arms: Plate fixation

SUMMARY:
Proximal forearm fractures comprise approximately 5% of all fractures, with olecranon fractures accounting for almost 20% of thes fractures. There is limited conclusive evidence regarding the optimal treatment and outcome of these fractures with only one prospective randomized trial (1992) in the literature comparing tension band wire and plate fixation for displaced olecranon fracture. Our trial includes all patients under the age of 75yrs presenting to the Edinburgh Orthopaedic Trauma Unit with an isolated olecranon fracture requiring operative intervention. Patients who consent to enrol in the trial will be randomised to operative fixation using one of two recognised fixation techniques - tension band wire fixation or plate fixation. Patients will be evaluated over a one year period following their surgery.

DETAILED DESCRIPTION:
Background

Proximal forearm fractures comprise approximately 5% of all fractures, whilst olecranon fractures account for almost 20% of fractures occurring around the elbow1. There is limited conclusive evidence regarding the epidemiology, optimal treatment and outcome of isolated olecranon fractures.

Patients with undisplaced olecranon fractures can be treated non-operatively2,3. The aims of treatment in displaced olecranon fractures are the restoration of function and stability to the elbow joint4. The technique employed should allow preservation and reconstruction of the articular surface with minimal associated complications. Tension-band wiring (TBW) is the most recognised and commonly used fixation method, although plate fixation and intramedullary screw fixation are noted alternatives2,4-10. Potential problems with the TBW technique are wound breakdown, infection, prominent metalwork, malunion and non-union2,4,7,11-13. Furthermore, plate fixation is considered to be superior in distal/comminuted/oblique fractures and fracture-dislocations, with superior fracture reduction and fixation results, as well as a lower rate of re-operation2,5,13,14. There is only one prospective randomized trial in the literature comparing TBW and plate fixation for displaced olecranon fracture13. The major conclusions from this study were:

* The functional outcome at six months was not significantly different in the two groups
* Post-operative loss of fracture reduction (53% vs 5%) and prominent symptomatic metalwork was more frequently observed after TBW

This study was performed in 1992 with less sophisticated plates when compared with the location specific plates currently available.

Research Aim

To determine if any difference exists in outcome (primary measure - DASH score) after one year between open reduction and internal fixation with tension band wiring AND plate and screw fixation for olecranon fractures.

Methodology

This trial involves identifying patients under the age of 75yrs (<75yrs) presenting to the Edinburgh Orthopaedic Trauma Unit with an isolated olecranon fracture requiring operative intervention. Patients who consent to enrol in the trial will be randomised to one of two recognised operative fixation techniques - tension band wire fixation or plate fixation. The trial will commence once ethical approval is granted by the Lothian Research Ethics Committee.

All statistical analysis was/will be performed by Dr Rob Elton. Prior to the study a power analysis determined the number of patients required in each trial. The primary outcome measure will be the DASH score, a continuous variable that follows a normal (Gaussian-shaped) distribution. This study is designed to determine a clinically relevant mean difference of 10 points between the two cohorts at one year after enrolment. A power analysis indicated that a total sample size of 50 (25 in each group) subjects will provide 80% statistical power to detect significant differences (0.05) in DASH scores, assuming an effect size of 0.8 (mean difference of 10 points, standard deviation of 12 points) using an unpaired t-test. To account for a possible loss to follow-up of up to 25%, we anticipate enrolling 35 subjects in each cohort for a total sample size of 70 subjects. A p value of < 0.05 was considered statistically significant.

All adult patients presenting to the Edinburgh Orthopaedic Trauma Unit with a fracture of the olecranon that satisfy the inclusion criteria will be invited to participate in our study. All adult patients with an olecranon fracture best treated operatively are eligible for enrolment in this study regardless of sex, race or ethnicity. Vulnerable populations will not be recruited.

A qualified member of the on-call team will introduce the study to the patient and initiate informed consent. If the patient agrees, a research fellow (Trauma and Orthopaedic StR3 level), not involved with the patient's care will review the study protocol in detail and address any questions the patient may have. If the patient is willing to participate, the research fellow will complete the informed consent. Patients will be given a copy of the consent form, and be informed that their participation is voluntary and that they can withdraw at any time during the study without detriment to their normal care in any way. Patients may take as long as they like to consider participation, provided that they still meet all the eligibility criteria documented above. Patients that are willing to participate in this study will get the same care of their fracture as patients that decide not to participate in the study.

On enrolment, a data collection form will be started with demographic and injury-related information collected. Prior to surgery, patients will be randomised (performed by Dr Rob Elton using closed opaque envelopes) into one of the two groups (tension band wire fixation or plate fixation). Following surgery, the post-operative assessment and course will be as per normal protocol for patients who are not in this study. Patients will be immobilised depending on fracture fixation during surgery and the decision will be made by the treating surgeon. Physiotherapy will be arranged when required

Follow-up All follow-up assessment will take place during follow-up visits initially with the treating consultant surgeon's team and a dedicated research physiotherapist. Radiographs and other diagnostic studies will be obtained at the discretion of the treating surgeon and will not differ from routine clinical care.

Follow-up assessment will be collected over a one year period (2 weeks, 6 weeks, 3 months, 6 months and one year). Routine follow-up in our institution for patients who have sustained an olecranon fracture that is managed operatively involves outpatient clinic reviews with radiographs at 2 weeks, 6 weeks, three months and six months. Therefore, one additional visit at 1 year is required for this study with no additional radiographs. Radiographs will only be performed at one year on clinical indication.

At each visit physical examination, treatment, complications and re-operation (e.g. hardware removal), for each patient will be recorded. A research physiotherapist, blinded to the treatment method by sticking plaster over the entry position, will undertake functional testing and assessment.

Outcome and statistical methods By statistically analysing the outcome scores in the two groups, I aim to better determine the optimal management of this fracture in this age group. Using univariate analysis and multivariate regression analysis I will determine significant (p<0.05) predictors of outcome in relation to functional outcome score (DASH at one year).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥16 years to <75yrs
2. Minimal/moderate fragmentation of the olecranon
3. Within two weeks of olecranon fracture

Exclusion Criteria:

1. Pregnant women with pre-determined treatment
2. Patients unable to give informed consent
3. Associated fractures to the coronoid, radial head and/or distal humerus
4. Associated ligamentous injury, dislocation or subluxation
5. Open fractures

Ages: 16 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2010-09; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
DASH | One year
  Patient rated outcome measure - DASH questionnaire at one year post injury/surgery.

SECONDARY OUTCOMES:
Mayo Elbow Performance Index (MEPI) | One year
  Completion of the Mayo Elbow Performance Index (MEPI), a physician rate scale of function will completed for all patients15. The MEPI is a validated hundred-point system based upon pain (forty five points), range of motion (twenty points), stability (ten points) and daily function (twenty five points). Categorical ratings are assigned as follows: ninety to one hundred points is rated excellent; seventy-five to eighty-nine, good; sixty to seventy-four, fair; and less than sixty points, poor.
Range of motion | One year
  Range of motion at the elbow and forearm: will be measured using a standard full circle goniometer. Flexion, extension, supination and prontation will be measured in triplicate and the mean recorded to minimise intra-observer bias
Pain | One year
  Pain assessment on an analogue scale 1-10.
Radiographic Assessment | Six months
  Radiographic assessment used standard anteroposterior (AP) and lateral radiographs of the elbow. Outcome will also be assessed in detail with regards to loss of fracture reduction, complications, union and the development of radiographic degenerative changes.
Time taken to return to activities | One year
  Time taken to return to activities of daily living/work/sport

CONTACTS AND LOCATIONS:
Overall Officials: Margaret M McQueen, MD, FRCSEd, Principal Investigator — Edinburgh Orthopaedic Trauma Unit
Locations (1):
- Edinburgh Orthopaedic Trauma Unit, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Peer reviewed publication - under review

REFERENCES:
- [Background] Newman SD, Mauffrey C, Krikler S. Olecranon fractures. Injury. 2009 Jun;40(6):575-81. doi: 10.1016/j.injury.2008.12.013. Epub 2009 Apr 23. PMID 19394931
- [Background] Veras Del Monte L, Sirera Vercher M, Busquets Net R, Castellanos Robles J, Carrera Calderer L, Mir Bullo X. Conservative treatment of displaced fractures of the olecranon in the elderly. Injury. 1999 Mar;30(2):105-10. doi: 10.1016/s0020-1383(98)00223-x. PMID 10476278
- [Background] Rommens PM, Kuchle R, Schneider RU, Reuter M. Olecranon fractures in adults: factors influencing outcome. Injury. 2004 Nov;35(11):1149-57. doi: 10.1016/j.injury.2003.12.002. PMID 15488508
- [Background] Fyfe IS, Mossad MM, Holdsworth BJ. Methods of fixation of olecranon fractures. An experimental mechanical study. J Bone Joint Surg Br. 1985 May;67(3):367-72. doi: 10.1302/0301-620X.67B3.3997942.
- [Background] Karlsson MK, Hasserius R, Karlsson C, Besjakov J, Josefsson PO. Fractures of the olecranon: a 15- to 25-year followup of 73 patients. Clin Orthop Relat Res. 2002 Oct;(403):205-12. PMID 12360028
- [Background] Chalidis BE, Sachinis NC, Samoladas EP, Dimitriou CG, Pournaras JD. Is tension band wiring technique the "gold standard" for the treatment of olecranon fractures? A long term functional outcome study. J Orthop Surg Res. 2008 Feb 22;3:9. doi: 10.1186/1749-799X-3-9. PMID 18294381
- [Background] Murphy DF, Greene WB, Gilbert JA, Dameron TB Jr. Displaced olecranon fractures in adults. Biomechanical analysis of fixation methods. Clin Orthop Relat Res. 1987 Nov;(224):210-4. PMID 3665242
- [Background] Murphy DF, Greene WB, Dameron TB Jr. Displaced olecranon fractures in adults. Clinical evaluation. Clin Orthop Relat Res. 1987 Nov;(224):215-23. PMID 3665243
- [Background] Gartsman GM, Sculco TP, Otis JC. Operative treatment of olecranon fractures. Excision or open reduction with internal fixation. J Bone Joint Surg Am. 1981 Jun;63(5):718-21. PMID 7240294
- [Background] Macko D, Szabo RM. Complications of tension-band wiring of olecranon fractures. J Bone Joint Surg Am. 1985 Dec;67(9):1396-401. PMID 3908460
- [Background] Hume MC, Wiss DA. Olecranon fractures. A clinical and radiographic comparison of tension band wiring and plate fixation. Clin Orthop Relat Res. 1992 Dec;(285):229-35. PMID 1446443
- [Background] Bailey CS, MacDermid J, Patterson SD, King GJ. Outcome of plate fixation of olecranon fractures. J Orthop Trauma. 2001 Nov;15(8):542-8. doi: 10.1097/00005131-200111000-00002. PMID 11733669
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720